CLINICAL TRIAL: NCT00687453
Title: The Utility of Insulin Glargine (Lantus) Compared to NPH in Ethnic Minority Type 2 Diabetic Subjects on Combination Insulin-Oral Agent Therapy
Brief Title: Insulin Glargine Versus Twice-Daily NPH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-02-519; U54RR014616 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glargine; Type 2 diabetes; Basal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glargine injected at bedtime (Experimental): Insulin glargine injected at bedtime
  Interventions: Drug: Insulin glargine at bedtime instead of NPH
- NPH insulin injected twice-daily (Active Comparator): NPH insulin injected twice-daily, before breakfast and at bedtime
  Interventions: Drug: NPH twice-daily

INTERVENTIONS:
Drug: Insulin glargine at bedtime instead of NPH — Insulin glargine at bedtime substituting for NPH insulin at bedtime
  Other Names: Trade name: Lantus
  Arms: Insulin glargine injected at bedtime
Drug: NPH twice-daily — Addition of morning NPH to bedtime NPH
  Other Names: (Generic)
  Arms: NPH insulin injected twice-daily

SUMMARY:
To compare the efficacy and safety of once-nightly insulin glargine versus twice-daily NPH insulin in ethnic minority type 2 diabetic patients inadequately treated with once-nightly NPH insulin alone.

DETAILED DESCRIPTION:
Insulin glargine has a longer action than compared to NPH insulin, but whether this results in improved control when compared to twice-daily NPH insulin is not known when used in low-income ethnic minority patients. This study investigates whether insulin glargine may be more or less effective and safe than twice-daily NPH insulin in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75
* Type 2 diabetes diagnosed for at least 1 year
* Inadequate glycemic control (hemoglobin A1c ≥ 7.5%) on stable and maximum-tolerated doses of a sulfonylurea, metformin and a thiazolidinedione, plus a single bedtime injection of NPH insulin
* Except for the subject's current bedtime NPH insulin, no other past history of chronic insulin use (other than treatment of gestational diabetes or hospitalizations of less than 1 week in duration)
* Average fasting plasma glucose level <130 mg/dL without fasting hypoglycemia
* Hemoglobin A1c between 7.5% and 12%
* Body mass index (BMI) between 20 and 40 kg/m2

Exclusion Criteria:

* History of confirmed (or clinical suspicion of ) type 1 diabetes
* Female subjects of childbearing potential who are sexually active and not using a reliable form of contraception.
* Current pregnancy or lactation.
* Subjects for whom intensive insulin therapy is contraindicated
* Subjects with advanced proliferative diabetic retinopathy
* Subjects who are unable to stay on a consistent daily meal schedule
* History of any clinically significant renal, hepatic, cardiovascular, neurological, endocrinological or other major systemic disease that, in the opinion of the investigator, may make implementation of the protocol or interpretation of the data difficult.
* Subjects who will likely require or initiate therapy with drugs which may interfere with glucose metabolism during the course of the study
* Subjects who are in another investigational study or have received another investigational medication within 30 days of study entry
* Subjects who are unable or unwilling to comply with all components of the study protocol, including contacting the investigators at specified times and attending all scheduled follow-up visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from Feb 2003 to Dec 2008. Subjects recruited from a diabetes specialty referral clinic, as well as from primary care clinics and through advertising in the South Los Angeles area.
Pre-assignment Details: Baseline run-in period to document baseline control and reinforce dietary/lifestyle principles.
  3 subjects not randomized due to protocol violations.
Groups:
- Insulin Glargine at Bedtime: Bedtime insulin glargine titrated to morning fasting glucose readings
- NPH Twice-daily: Morning and bedtime NPH insulin titrated to pre-supper and fasting glucose readings, respectively
Period: Overall Study
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Started | 11 | 13
Completed | 8 | 7
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (7.0) | 54.6 (7.6) | 55.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 9.1 (1.4) | 9.5 (1.2) | 9.3 (1.3)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 146 (75) | 145 (34) | 146 (56)
Diabetes Duration [Mean (Standard Deviation); unit: Years] | 9.4 (3.5) | 11.5 (4.0) | 10.6 (3.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (4.1) | 33.5 (6.6) | 31.8 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c Change From Baseline
Time Frame: Baseline to 6 months
Population: ITT (LOCF)
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
Percent glycated hemoglobin | -0.8 (0.9) | -1.0 (1.2)

2. Secondary Outcome: Frequency of Pre-supper Glucose Readings 130 mg/dL or Less, Change From Baseline
Time Frame: 6 months
Population: ITT (LOCF)
Measure: Mean (Standard Deviation); unit: % of readings, change from baseline
Groups:
- Insulin Glargine at Bedtime: Insulin glargine at bedtime instead of NPH: Insulin glargine at bedtime substituting for NPH insulin at bedtime
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
% of readings, change from baseline | 38.0 (30.1) | 7.5 (22.6)

3. Secondary Outcome: Frequency of Total Hypoglycemic Reactions
Time Frame: 6 months
Population: ITT (LOCF)
Measure: Number; unit: Events
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
Events | 55 | 28

4. Secondary Outcome: Frequency of Severe Hypoglycemic Reactions
Time Frame: 6 months
Population: ITT (LOCF)
Measure: Number; unit: Events
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
Events | 0 | 0

5. Secondary Outcome: Body Mass Index Change From Baseline
Time Frame: Baseline and 6 months
Population: ITT (LOCF)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Insulin Glargine Injected at Bedtime | NPH Insulin Injected Twice-daily
Number analyzed (Participants) | 11 | 13
kg/m^2 | 0.2 (1.0) | 0.3 (1.2)

6. Secondary Outcome: Total Daily Insulin Dose
Time Frame: Baseline and 6 months
Population: ITT (LOCF)
Measure: Mean (Standard Deviation); unit: Units per day, change from baseline
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
Units per day, change from baseline | -0.1 (14.4) | 20.5 (9.8)

7. Secondary Outcome: Any Adverse Event Other Than Hypoglycemia
Time Frame: 6 months
Measure: Number; unit: Events
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
Number analyzed (Participants) | 11 | 13
Events | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Insulin Glargine at Bedtime | NPH Twice-daily
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 8/11 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine at Bedtime (N=11) | NPH Twice-daily (N=13)
Symptomatic Hypoglycemia (Endocrine disorders) | 8 (55) | 5 (28) — Classic symptoms of hypoglycemia, relieved by carbohydrate ingestion, with or without a corroborating self-monitored glucose reading
Peripheral Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to smaller than anticipated enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes